CLINICAL TRIAL: NCT00175006
Title: A Study to Assess a Direct Physical Measurement Method for Evaluation of Tophus Nodules in Subjects With Gout.
Brief Title: Validation Study of Physical Measurement of Tophi
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP, Clinical Science, Takeda Global Research & Development Center, Inc.
Other Study IDs: C02-019; U1111-1114-1944 (Registry Identifier: WHO)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2009-07-16 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Gout
Keywords: Hyperuricemia; Tophi; Tophus; Drug Therapy
MeSH Terms: conditions — Gout; Hyperuricemia

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: None Retained — None taken or retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tophi Participants
  Interventions: Other: Measurement of Tophi to validate procedure

INTERVENTIONS:
Other: Measurement of Tophi to validate procedure — Intra- and Inter-rater Reproducibility measurements of the area (in mm2) of each tophus nodule.

SUMMARY:
The purpose of this study is to determine the inter- and intra-rater reproducibility of direct physical measurement of tophus nodules in subjects with gout.

DETAILED DESCRIPTION:
Gout is a chronic urate crystal deposition disorder. Left untreated, gout may result in progressive disease characterized by joint and bone destruction from tophaceous deposits and renal impairment due to gouty nephropathy. Hyperuricemia, defined as a serum urate concentration greater than 7.0 milligrams per deciliter (mg/dL), is the underlying metabolic aberration leading to urate crystal deposition in gout. Gout has several clinical presentations, including: recurrent acute attacks of inflammatory arthritis; deposition of monosodium urate monohydrate crystals in joints, bones and even parenchymal organs (tophaceous gout); renal impairment; and uric acid nephrolithiasis.1 As serum urate levels increase beyond greater than 7.0 mg/dL, the risks for gouty arthritis or for renal calculi increase.

Febuxostat is a 2-aryl-thiazole derivative chemically engineered as a novel xanthine oxidase/dehydrogenase inhibitor. Febuxostat is being developed as an orally administered agent for the management of hyperuricemia in patients with gout.

Subjects with palpable tophi >10 millimeters (mm) in length and width and as round as possible will have the tophus measured on two separate visits by two different raters to assess the inter- and intra-rater reproducibility of direct physical measurement.

ELIGIBILITY:
Inclusion Criteria:

* Must have at least 1 palpable gouty tophus nodule in the foot/ankle, hand/wrist, or elbow, confirmed as gouty by prior diagnosis according to ACR criteria.
* The tophus must be solid, round, non-tender, intact, and larger than 10mm in both length and width.
* Joints nearest and immediately adjacent to the selected tophus must not be acutely inflamed.
* Must be on stable treatment for gout with no medication changes in the past 30 days.

Exclusion Criteria:

* Must be able to return to the clinical site within 10 days.
* Must not have allergy to ink.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with palpable tophi >10mm in length and width and as round as possible will have the tophus measured on two separate visits by two different raters to assess the inter- and intra-rater reproducibility of direct physical measurement.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2002-11; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda

REFERENCES:
- [Result] Schumacher HR Jr, Becker MA, Palo WA, Streit J, MacDonald PA, Joseph-Ridge N. Tophaceous gout: quantitative evaluation by direct physical measurement. J Rheumatol. 2005 Dec;32(12):2368-72. PMID 16331766
- See also: Uloric Package Insert — http://general.takedapharm.com/content/file.aspx?applicationcode=6C7C39D8-5D09-453B-BF30-696A4AB88E62&fileTypeCode=ULORICPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 2 study sites in the United States from 19 November 2002 to 09 January 2003.
Groups:
- Tophi Participants: Participants with palpable tophi >10 millimeters (mm) in length and width and as round as possible measured on two separate visits by two different raters.
Period: Overall Study
Arm/Group | Tophi Participants
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tophi Participants
Number analyzed (Participants) | 13
Age Continuous [Mean (Standard Deviation); unit: years] | 60.5 (14.1)
Age, Customized [Number; unit: participants]
  18 years to 35 years | 0
  36 years to 50 years | 2
  51 years to 65 years | 6
  66 years to 85 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 11
Race/Ethnicity, Customized [Number; unit: participants]
  White | 5
  Black or African American | 7
  Asian | 1

OUTCOME MEASURES:

1. Primary Outcome: Average Percent Difference in Area Between Visits
Description: The rater measured length and width (mm) of the tophus at 2 visits separated by no more than 10 days. Area of the tophus was summarized using average percent difference, calculated as absolute difference of Visits 1 and 2 divided by the average of Visits 1 and 2 for the same tophus, pooled across raters.
Time Frame: Visit 1 (Day 1) and Visit 2 (Days 6-11)
Population: Measurements of 52 tophi were obtained at 2 separate visits separated by no more than 10 days from the 13 subjects enrolled. Change in tophus size over 10 days was not expected.
Measure: Mean (Standard Deviation); unit: mm²
Arm/Group | Tophi Participants
Number analyzed (Participants) | 13
mm²
  Average Percent Difference | 29 (33)

2. Primary Outcome: Average Percent Difference in Area Between Raters
Description: Each rater measured length and width (mm) of the tophus at 2 visits separated by no more than 10 days. Area of the tophus was summarized using the average percent difference, calculated as the absolute difference of Raters 1 and 2 divided by the average of Raters 1 and 2 for the same tophus, pooled across visits.
Time Frame: Visit 1 (Day 1 ) and Visit 2 (Day 6-11)
Population: Measurements of 52 tophi were obtained at 2 separate visits separated by no more than 10 days from the 13 subjects enrolled.
Measure: Mean (Standard Deviation); unit: mm²
Arm/Group | Tophi Participants
Number analyzed (Participants) | 13
mm²
  Average Percent Difference | 32 (27)

ADVERSE EVENTS:
Arm/Group | Tophi Participants
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.